CLINICAL TRIAL: NCT05817708
Title: A Dose Selection Phase 1 Study Evaluating the Safety and Tolerability of Silmitasertib
Brief Title: A Study of Silmitasertib (CX-4945) in Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Senhwa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX4945-AV04-phase I
Record Dates: First submitted 2023-01-30; First posted 2023-04-18 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — silmitasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CX-4945 200mg QD (Experimental): CX-4945 will be administered at 200mg QD for continuously 5 days.
  Interventions: Drug: CX-4945
- CX-4945 200mg BID (Experimental): CX-4945 will be administered at 200mg BID for continuously 5 days.
  Interventions: Drug: CX-4945
- CX-4945 400mg BID (Experimental): CX-4945 will be administered at 400mg BID for continuously 5 days.
  Interventions: Drug: CX-4945

INTERVENTIONS:
Drug: CX-4945 — Drug: CX-4945
  Silmitasertib, orally, once or twice daily for 5 days.
  Other Name: Silmitasertib
  Other Names: Silmitasertib

SUMMARY:
This is a Phase I single center, open-label, parallel design in 30 subjects to evaluate safety and tolerability of CX-4945 200mg QD, 200 mg BID and 400mg BID doses (10 subjects in each regimen) for continuously 5 days in healthy subjects for dose selection.

DETAILED DESCRIPTION:
COVID-19 is characterized by SARS-CoV-2 induced up-regulation of host protein kinase CK2 that catalyzes phosphorylation of many proteins, modulating their activities in cellular processes. CX-4945 demonstrated anti-viral efficacy in COVID-19 in vitro studies. In CX4945-AV01-IIT(IND 152726), CX-4945 was a safe treatment at 1000 mg BID regimen supported by the fact of no occurrence of treatment related Grade ≥ 3 AE, death or SUSAR. There were approximately 50 % of patients who experienced gastrointestinal disorders of grade 1-2. In CX4945-AV01-IIT, an out-patient study, there were 50% experienced gastrointestinal disorders. To further evaluate the safety and tolerability of CX-4945, this phase 1 study will use lower doses and subjects will be close-monitored to evaluate the safety.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects 20to 55 years of age, inclusive, at screening
2. Body mass index (BMI)within the range of 18.0 to 30.0 kg/m2, inclusive, and a minimum weight of 50.0 kg at screening
3. Subjects who are of reproductive potential agreed to remain abstinent or use (or have their partner use) an acceptable method of birth control (intrauterine device, hormonal contraception, vasectomy or condom) from screening until at least 2 weeks after the last study drug administration.
4. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, and electrocardiogram;
5. Subject with acceptable hematology, biochemistry and urinalysis during screening period.
6. Subject is willing and able to comply with study procedures and sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and from screening until at least 2 weeks after the last study drug administration. Should a man father a child, or a woman become pregnant or suspect she is pregnant while participating in this study, he or she should inform the treating physician immediately.
2. Active or uncontrolled infections such asCOVID-19, HIV or with serious illnesses or medical conditions which would not permit the subject to receive study treatment.
3. Subject has received any prescription of drug within 3 days prior to study enrollment.
4. Subject has drug abuse history.
5. Any active or recurring clinically significant hepatic disease including HBV and HCV.
6. Subject has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of investigational product.
7. Any other medical reason as determined by the investigator.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ding Huang, PhD, Study Director — Senhwa Biosciences
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from healthy subjects at Taipei Medical University Hospital between November 2022 and December 2022. The first participant was enrolled on November 28th, 2022, and the last was enrolled in 28th December 2022.
Pre-assignment Details: 30 enrolled participants met inclusion criteria and were randomized.
Groups:
- CX-4945 200mg QD: CX-4945 will be administered at 200mg QD for continuously 5 days.
  CX-4945: Drug: CX-4945
  Silmitasertib, orally, once or twice daily for 5 days.
  Other Name: Silmitasertib
- CX-4945 200mg BID: CX-4945 will be administered at 200mg BID for continuously 5 days.
  CX-4945: Drug: CX-4945
  Silmitasertib, orally, once or twice daily for 5 days.
  Other Name: Silmitasertib
- CX-4945 400mg BID: CX-4945 will be administered at 400mg BID for continuously 5 days.
  CX-4945: Drug: CX-4945
  Silmitasertib, orally, once or twice daily for 5 days.
  Other Name: Silmitasertib
Period: Overall Study
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- CX-4945 200mg QD: CX-4945 was administered at 200mg QD for continuously 5 days.
- CX-4945 200mg BID: CX-4945 was administered at 200mg BID for continuously 5 days.
- CX-4945 400mg BID: CX-4945 was administered at 400mg BID for continuously 5 days.
- Total: Total of all reporting groups
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Median (Full Range); unit: years] | 33.5 [27 to 38] | 32 [21 to 46] | 37.5 [29 to 45] | 33.5 [21 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 10
  Male | 5 | 7 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 10 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 10 | 10 | 10 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAT)
Description: Evaluate the number adverse events occurring from Day 1 to Day 5 as characterized by type, frequency, severity [as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE] version 5.0], timing, seriousness, and relationship to study therapy after administration of 200mg QD, 200mg BID and 400mg BID for continuously 5 days to healthy subjects.
Time Frame: Day 1 to Day 5
Population: Treatment-Emergent Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
Participants | 1 | 3 | 7

2. Secondary Outcome: Evaluate Changes in Blood Chemistry.
Description: Changes ALP in blood chemistry assessment from Day 1(Baseline) to Day 6 morning.
Time Frame: Day 1 to Day 6
Population: Day 6 (EOT) - Change from Baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
U/L | -2.1 (5.78) | -0.3 (6.62) | 3.4 (2.84)

3. Secondary Outcome: Evaluate Changes in Blood Chemistry.
Description: Changes AST in blood chemistry assessment from Day 1(Baseline) to Day 6 morning.
Time Frame: Day 1 to Day 6
Population: Day 6 (EOT) - Change from Baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
U/L | -3.9 (5.11) | -2.4 (3.72) | 0.1 (3.35)

4. Secondary Outcome: To Evaluate Changes in Blood Chemistry.
Description: Changes ALT in blood chemistry assessment from Day 1(Baseline) to Day 6 morning.
Time Frame: Day 1 to Day 6
Population: Day 6 (EOT) - Change from Baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
U/L | -4.0 (6.15) | -1.4 (5.19) | 0.9 (4.77)

5. Secondary Outcome: To Evaluate Changes in Blood Chemistry.
Description: Changes LDH in blood chemistry assessment from Day 1(Baseline) to Day 6 morning.
Time Frame: Day 1 to Day 6
Population: Day 6 (EOT) - Change from Baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
U/L | -17.0 (17.17) | -26.2 (10.75) | -28.2 (14.33)

6. Secondary Outcome: To Evaluate Changes in Blood Chemistry.
Description: Changes CPK in blood chemistry assessment from Day 1(Baseline) to Day 6 morning.
Time Frame: Day 1 to Day 6
Population: Day 6 (EOT) - Change from Baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
U/L | -24.3 (19.35) | -54.0 (63.71) | -65.1 (71.37)

7. Secondary Outcome: To Evaluate Changes in Blood Chemistry.
Description: Changes CRP in blood chemistry assessment from Day 1(Baseline) to Day 6 morning.
Time Frame: Day 1 to Day 6
Population: Day 6 (EOT) - Change from Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
mg/dL | 0.003 (0.1341) | -0.071 (0.2497) | 0.002 (0.0447)

8. Secondary Outcome: Number of Participants Evaluated as Having Abnormalities (CS or NCS) in Their ECG
Description: ECG assessments were done during Screening, Day 1, Day 3, Day 5, and Day 6. A 12-lead ECG was performed at baseline (Day1), Day 3, Day 5, and Day 6 and categorized as normal, abnormal and not clinically significant (abnormal NCS) or abnormal and clinically significant (abnormal CS).
Time Frame: Screening, Day 1, Day 3, Day 5, and Day 6
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | CX-4945 200mg QD | CX-4945 200mg BID | CX-4945 400mg BID
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Screening | 7 | 6 | 6
  Day 1 (Baseline) | 3 | 4 | 8
  Day 3 | 7 | 9 | 6
  Day 5 | 5 | 6 | 7
  Day 6 | 6 | 6 | 6

ADVERSE EVENTS:
Time Frame: from Day 1 to Day 6
Description: Adverse Events experienced by patients from randomization(Day 1) to Day 6 (including vital signs, physical findings, clinical laboratory, and ECG results) as characterized by type, frequency, severity (as graded by Common Terminology Criteria for Adverse Events (CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Arm/Group | CX-4945 200mg BID | CX-4945 200mg QD | CX-4945 400mg BID
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 3/10 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CX-4945 200mg BID (N=10) | CX-4945 200mg QD (N=10) | CX-4945 400mg BID (N=10)
Dirrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
C-reactive protein abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT05817708/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT05817708/SAP_001.pdf